CLINICAL TRIAL: NCT02521714
Title: A Phase 1, Open-label, Randomized, Three-period, Two-way Crossover Study in Healthy Subjects to Evaluate the Bioavailability of a Test Lenalidomide Oral Suspension Relative to the Reference Capsule Formulation and to Assess the Effect of Food on the Bioavailability of Lenalidomide From the Oral Suspension
Brief Title: Study to Evaluatethe Bioavailability and Food Effect Lenalidomide as an Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CC-5013-CP-013
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Revlimid; lenalidomide; bioavailability; healthy volunteers; food effect; pharmacokinetics
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: 25mg capsule -under fasted condition (Experimental): Single oral dose of 25mg lenalidomide (reference formulation, 1 x 25mg capsule) under fasted condition.
  Interventions: Drug: Lenalidomide
- Treatment B: 25mg oral suspension - under fasted condition (Experimental): Single oral dose of 25mg lenalidomide (test formulation, 2.5mL oral suspension) under fasted condition.
  Interventions: Drug: Lenalidomide
- Treatment C: 25mg oral suspension -under fed condition (Experimental): Single oral dose of 25mg lenalidomide (test formulation, 2.5mL oral suspension) under fed condition.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid®

SUMMARY:
This study will evaluate the amount of drug that reaches the circulation when a subject takes the test (liquid) formulation compared to the reference (capsule) formulation. The study will also examine the effect of a high fat meal on the levels of drug in blood.

DETAILED DESCRIPTION:
This is a phase 1, open-label, randomized, three-period, two-way crossover study in healthy subjects. The study will consist of a screening phase, a baseline phase, three treatment periods, and a follow-up phone call. Each period will be two days in duration (Day 1 through Day 2) for dosing and sample collection. There will be a minimum of four days washout between doses.

Within no more than 21 days (Day -21) and no less than two days (Day -2) prior to the start of Period 1, subjects will undergo routine screening procedures including physical examination (PE), 12-lead electrocardiogram (ECG), vital signs, clinical laboratory safety tests (serum chemistry, hematology, and urinalysis), serology screen, and drug/alcohol screen.

Eligible subjects will be admitted into the study center on Day -1 of Period 1 for baseline assessments. During each period, subjects will receive a single 25 mg oral dose of lenalidomide on Day 1 according to the assigned treatment sequence. Serial blood sampling for the determination of lenalidomide concentrations in plasma will be performed for 24 hours post dose, and safety will be evaluated. Subjects will be domiciled at the study center from Day 1 of Period 1 through Day 2 of Period 3, including the 4 day washout between each dose of IP. All subjects will be discharged from the study center on Day 2 of Period 3 following completion of required study procedures.

A follow-up phone call will occur approximately four days (±2 days) after discharge from the study center.

The study will be conducted in compliance with International Conference on Harmonisation (ICH) Good Clinical Practices (GCPs).

ELIGIBILITY:
Inclusion Criteria:

- Subjects must satisfy the following criteria to be enrolled in the study:

1. Males and females (of non-childbearing potential ) from any race and 18 years of age to 65 years of age at the time of signing the informed consent document.
2. Subject must understand and voluntarily sign an informed consent prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules
5. Male subjects

   * Must agree to practice complete abstinence (True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [eg, calendar, ovulation, symptothermal or, post ovulation methods] and withdrawal are not acceptable methods of contraception.) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential (FCBP) while taking lenalidomide, during dose interruptions, and for at least 28 days after the last dose of lenalidomide, even if he has undergone a successful vasectomy.
   * Must not donate semen or sperm while receiving lenalidomide, during dose interruptions, and for at least 28 days after the last dose of lenalidomide.
6. Counseling about pregnancy precautions and the potential risks of fetal exposure must be conducted as described in the Lenalidomide Pregnancy Prevention Plan.
7. Must have a body mass index (BMI) between 18 and 33 kg/m2 (inclusive).
8. Clinical laboratory tests must be within normal limits or considered not clinically significant by the investigator.
9. Must have confirmation of normal renal function.
10. Must be afebrile with supine systolic blood pressure: 90 to 140 mmHg, supine diastolic blood pressure: 50 to 90 mmHg, and pulse rate: 40 to 110 beats per minute at the screening visit. Vital signs may be repeated up to three times to determine eligibility.
11. Must have a normal or clinically acceptable 12-lead electrocardiogram, with a QTcF value ≤ 450 msec for male subjects or ≤ 470 msec for female subjects.

Exclusion Criteria:

- The presence of any of the following will exclude a subject from enrollment:

1. Any significant medical condition (e.g., renal insufficiency), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Used any prescribed systemic or topical medication within 30 days of the first dose administration, unless Sponsor agreement is obtained.
5. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless Sponsor agreement is obtained.
6. Has any surgical or medical conditions (excluding appendectomy) possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure, cholecystectomy.
7. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before the first dose administration , or positive alcohol screen.
10. Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb), or have a positive result to the test for HIV antibodies at Screening.
11. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2015-08-14 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUCt | approximately 11 days
  Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration
Pharmacokinetics - AUC∞ | approximately 11 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - Cmax | approximately 11 days
  Maximum observed plasma concentration
Pharmacokinetics - Tmax | approximately 11 days
  Time to maximum plasma concentration
Pharmacokinetics - T1/2 | approximately 11 days
  Terminal phase half-life in plasma
Pharmacokinetics - CL/F | approximately 11 days
  Apparent total clearance when dosed orally
Pharmacokinetics - Vz/F | approximately 11 days
  Apparent volume of distribution when dosed orally

SECONDARY OUTCOMES:
Adverse Events (AEs) | up to 5 weeks
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ramirez-Valle, MD, PhD, Study Director — Celgene Corporation
Locations (1):
- Covance-Daytona Beach, Daytona Beach, Florida, United States